CLINICAL TRIAL: NCT06853327
Title: Timing of Oral Ketorolac for Pain Reduction in IUD Insertion: A Double-Blind Randomized Controlled Trial
Brief Title: Oral Ketorolac for IUD Pain Reduction
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-2276
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: IUD Insertion Pain
Keywords: IUD; Intrauterine Device; Ketorolac; IUD pain; NSAID; Non-steroidal Anti-Inflammatory Drug; VAS; PASS
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- K2 - Ketorolac 2-hour (Active Comparator): Receives Ketorolac 20mg PO at 2 hours prior and placebo at 1 hour prior to IUD
  Interventions: Drug: Ketorolac; Drug: Placebo
- K1 - Ketorolac 1-hour (Active Comparator): Receives placebo at 2 hours and Ketorolac 20mg PO at 1 hour prior to IUD
  Interventions: Drug: Ketorolac; Drug: Placebo
- K0 - Placebo control (Placebo Comparator): Receives placebo at 2 hours and at 1 hour prior to IUD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — The experimental condition to be examined by this study is the timing of administration of ketorolac prior to IUD insertion. Ketorolac 20mg PO has proven beneficial at certain timepoints during IUD insertion in prior studies, but pharmacokinetics indicate that it could require more time until peak analgesia.
  Other Names: Toradol
  Arms: K1 - Ketorolac 1-hour; K2 - Ketorolac 2-hour
Drug: Placebo — Placebo will be used to control the timing of administration and be used to compare ketorolac to baseline standard pain control regimens

SUMMARY:
To determine if oral ketorolac given at different timepoints prior to intrauterine device (IUD) insertion influences pain experienced during this procedure.

DETAILED DESCRIPTION:
This is a single-site prospective interventional randomized controlled trial to examine the timing of administration of ketorolac for IUD pain control. 108 patients will be recruited to the study and they will be randomized into three study arms in a 1:1:1 ratio. Information including demographics, medical history, and obstetric history will be collected during enrollment. Patients will arrive 3 hours prior to their IUD appointment. Study group "K2" will receive ketorolac 20mg per os (PO) at 2 hours prior to IUD insertion, then they will receive a placebo pill at 1 hour prior to IUD insertion. In contrast, study group "K1" will receive the inverse: they will be given a placebo pill at 2 hours prior to IUD insertion, then they will receive ketorolac 20mg PO at 1 hour prior to IUD insertion. Study group "K0" will receive placebo pills at both timepoints. The patients will then receive a standard IUD insertion by an OBGYN physician. Both patients and providers will be blinded to the study medications received. The standard pain control regimen for IUD insertion includes offering vaginal lidocaine gel self-administered 5 minutes prior to IUD insertion as well as offering lidocaine paracervical block (PCB). All patients will be offered these standard pain control methods including the "K0" group. Patients may utilize one, both, or neither of these offered interventions in addition to the randomized study medication. During the IUD insertion, pain scores at 7 different timepoints will be measured via a visual analog scale (VAS). The VAS is a 100mm visual tool that allows patients to rate the pain they are experiencing at each time interval. The 7 timepoints include: pre-procedure, tenaculum placement, block injection, uterine sounding, IUD deployment, overall (measured immediately post-procedure), and 10 minutes post-procedure. Information on Patient Acceptable Symptom State (PASS) and patient satisfaction will be collected during their appointment. After the 10-minute post-procedure VAS score and questionnaire, patients will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to consent
* Desires IUD insertion

Exclusion Criteria:

* IUD placement under sedation or oral anxiolytic
* IUD replacement (removal with insertion)
* Daily narcotic or NSAID use
* Contraindications to IUD placement
* Current: pregnancy, genital/pelvic infection
* Lifetime history: uterine anomaly, pelvic inflammatory disease, allergy to levonorgestrel or copper
* Contraindications to ketorolac
* Current: weight under 50 kilograms
* Lifetime history: allergy to NSAIDs, liver disease, renal disease, peptic ulcer disease, cerebrovascular bleeding, gastrointestinal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in mean VAS pain scores between study arms at 7 timepoints during and after IUD insertion | All VAS pain scores will be measured during their IUD appointment. 5 timepoints will be measured during IUD insertion (~10 total minutes), 1 immediately after the procedure, 1 ten minutes afterwards
  To compare the mean VAS pain scores between study arms (K2 vs K1 vs K0) at each timepoint during and after IUD insertion (pre-procedure, tenaculum placement, PCB injection, uterine sounding, IUD deployment, overall (measured immediately post-procedure), and 10 minutes post-procedure). To assess VAS scores, a 100mm ruler will be presented to the patient at the listed timepoints. The patient will adjust a slider on the ruler to correspond to their pain level, with 0mm representing no pain and 100mm representing worst possible pain. The VAS scores will be reported as means and compared via repeated measure ANOVA test yielding confidence intervals and p-values and to assess for significance.

SECONDARY OUTCOMES:
Difference in mean VAS pain scores between study arms at 7 timepoints during and after IUD insertion, controlling for parity | Parity is recorded during intake 1 week prior to IUD. VAS pain scores will be measured during their IUD appointment. 5 timepoints will be measured during IUD insertion (~10 total minutes), 1 immediately after the procedure, 1 ten minutes afterwards
  To compare the mean VAS pain scores between study arms (K2 vs K1 vs K0) at each timepoint during and after IUD insertion (pre-procedure, tenaculum placement, PCB injection, uterine sounding, IUD deployment, overall (measured immediately post-procedure), and 10 minutes post-procedure) with respect to parity. To assess VAS scores, a 100mm ruler will be presented to the patient at the listed timepoints. The patient will adjust a slider on the ruler to correspond to their pain level, with 0mm representing no pain and 100mm representing worst possible pain. This will determine if nulliparous patients experienced more pain relief with different timings of ketorolac administration. The VAS scores for nulliparous and multiparous patients will be reported as means and compared via repeated measure ANOVA test with interaction term yielding confidence intervals and p-values to assess for significance.
Difference in rate of "severe pain" (VAS pain scores 70-100mm) between study arms at 7 timepoints during and after IUD insertion | All VAS pain scores will be measured during their IUD appointment. 5 timepoints will be measured during IUD insertion (~10 total minutes), 1 immediately after the procedure, 1 ten minutes afterwards
  To compare the rate of "severe pain" (VAS pain scores 70-100mm) between study arms (K2 vs K1 vs K0) at each timepoint during and after IUD insertion (pre-procedure, tenaculum placement, PCB injection, uterine sounding, IUD deployment, overall (measured immediately post-procedure), and 10 minutes post-procedure). To assess VAS scores, a 100mm ruler will be presented to the patient at the listed timepoints. The patient will adjust a slider on the ruler to correspond to their pain level, with 0mm representing no pain and 100mm representing worst possible pain. The rate of severe pain will be reported as percentage of patients and will be compared via chi-square test yielding confidence intervals and p-values to assess for significance.
Difference in rate of change of VAS pain scores between study arms at 7 timepoints during and after IUD insertion | All VAS pain scores will be measured during their IUD appointment. 5 timepoints will be measured during IUD insertion (~10 total minutes), 1 immediately after the procedure, 1 ten minutes afterwards
  To compare the rate of change of VAS pain scores between study arms (K2 vs K1 vs K0) at each timepoint during and after IUD insertion (pre-procedure, tenaculum placement, PCB injection, uterine sounding, IUD deployment, overall (measured immediately post-procedure), and 10 minutes post-procedure). To assess VAS scores, a 100mm ruler will be presented to the patient at the listed timepoints. The patient will adjust a slider on the ruler to correspond to their pain level, with 0mm representing no pain and 100mm representing worst possible pain. The pain scores will be plotted at the listed 7 timepoints and a generalized estimating equation will be used to assess the change in slope from timepoint to timepoint. The change in slope will be reported as means and compared between study arms via repeated measure ANOVA test yielding confidence intervals and p-values and to assess for significance.
Difference in rate of acceptable pain levels between study arms at 7 timepoints during and after IUD insertion | All PASS responses will be measured during their IUD appointment. 5 timepoints will be measured during IUD insertion (~10 total minutes), 1 immediately after the procedure, 1 ten minutes afterwards
  To compare the rate of acceptable pain levels (Patient Acceptable Symptom State (PASS) binary yes/no variable) between study arms (K2 vs K1 vs K0) at each timepoint during and after IUD insertion (pre-procedure, tenaculum placement, PCB injection, uterine sounding, IUD deployment, overall (measured immediately post-procedure), and 10 minutes post-procedure). To assess PASS, the patient will be asked "Do you consider your current pain level acceptable?" at the listed timepoints. The rate of acceptable pain levels will be reported as percentage of patients and will be compared via chi-square test yielding confidence intervals and p-values to assess for significance.

CONTACTS AND LOCATIONS:
Overall Officials: Amy G Bryant, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina - Hillsborough Campus, Hillsborough, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: beginning 9 and continuing for 36 months after publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.
URL: https://research.unc.edu/clinical-research-compliance/clinicaltrials-gov/icmje-data-sharing-statement-guidance/

REFERENCES:
- [Background] Crawford M, Davy S, Book N, Elliott JO, Arora A. Oral Ketorolac for Pain Relief During Intrauterine Device Insertion: A Double-Blinded Randomized Controlled Trial. J Obstet Gynaecol Can. 2017 Dec;39(12):1143-1149. doi: 10.1016/j.jogc.2017.05.014. Epub 2017 Aug 18. PMID 28826645
- [Background] Ngo LL, Ward KK, Mody SK. Ketorolac for Pain Control With Intrauterine Device Placement: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):29-36. doi: 10.1097/AOG.0000000000000912. PMID 26241253
- [Background] de Oliveira ECF, Baeta T, Brant APC, Silva-Filho A, Rocha ALL. Use of naproxen versus intracervical block for pain control during the 52-mg levonorgestrel-releasing intrauterine system insertion in young women: a multivariate analysis of a randomized controlled trial. BMC Womens Health. 2021 Oct 29;21(1):377. doi: 10.1186/s12905-021-01521-z. PMID 34715839
- [Background] Ngo LL, Braaten KP, Eichen E, Fortin J, Maurer R, Goldberg AB. Naproxen Sodium for Pain Control With Intrauterine Device Insertion: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1306-1313. doi: 10.1097/AOG.0000000000001746. PMID 27824753
- [Background] Bednarek PH, Creinin MD, Reeves MF, Cwiak C, Espey E, Jensen JT; Post-Aspiration IUD Randomization (PAIR) Study Trial Group. Prophylactic ibuprofen does not improve pain with IUD insertion: a randomized trial. Contraception. 2015 Mar;91(3):193-7. doi: 10.1016/j.contraception.2014.11.012. Epub 2014 Nov 25. PMID 25487172
- [Background] Reeves JA, Zapata LB, Curtis KM, Whiteman MK. Intrauterine Device Training, Attitudes, and Practices Among U.S. Health Care Providers: Findings from a Nationwide Survey. Womens Health Issues. 2023 Jan-Feb;33(1):45-53. doi: 10.1016/j.whi.2022.08.002. Epub 2022 Sep 16. PMID 36123229
- [Background] Akintomide H, Brima N, Sewell RD, Stephenson JM. Patients' experiences and providers' observations on pain during intrauterine device insertion. Eur J Contracept Reprod Health Care. 2015;20(4):319-26. doi: 10.3109/13625187.2015.1031885. Epub 2015 Apr 10. PMID 25857221
- [Background] Rahman M, King C, Saikaly R, Sosa M, Sibaja K, Tran B, Tran S, Morello P, Yeon Seo S, Yeon Seo Y, Jacobs RJ. Differing Approaches to Pain Management for Intrauterine Device Insertion and Maintenance: A Scoping Review. Cureus. 2024 Mar 8;16(3):e55785. doi: 10.7759/cureus.55785. eCollection 2024 Mar. PMID 38586685